CLINICAL TRIAL: NCT07232589
Title: A Study to Evaluate the Effect of Multiple Oral Doses of Diltiazem on the Single-Dose Pharmacokinetics of Nemtabrutinib in Healthy Participants.
Brief Title: A Study of the Effect of Diltiazem on the Plasma Levels of Nemtabrutinib (MK-1026-022)
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Basic Science
Other Study IDs: 1026-022; MK-1026-022 (Other: MSD)
Record Dates: First submitted 2025-11-14; First posted 2025-11-18 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Healthy
MeSH Terms: interventions — ARQ531; Diltiazem

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Period 1: Nemtabrutinib (Experimental): Participants will receive nemtabrutinib followed by a protocol specified wash-out period.
  Interventions: Drug: Nemtabrutinib
- Period 2: Diltiazem + Nemtabrutinib (Experimental): Participants will receive diltiazem plus nemtabrutinib.
  Interventions: Drug: Nemtabrutinib; Drug: Diltiazem

INTERVENTIONS:
Drug: Nemtabrutinib — Oral administration
  Other Names: MK-1026; ARQ 531
Drug: Diltiazem — Oral administration
  Arms: Period 2: Diltiazem + Nemtabrutinib

SUMMARY:
The goal of the study is to learn what happens to levels of nemtabrutinib (MK-1026) in a healthy person's body over time. Researchers will compare what happens to nemtabrutinib in the body when it is given with or without another medicine called diltiazem.

ELIGIBILITY:
Inclusion Criteria:

* Be in good health
* BMI between 18.5 and 32 kg/m2, inclusive

Exclusion Criteria:

* History of clinically significant endocrine, gastrointestinal, cardiovascular, hematological (history of a bleeding disorder, abnormal bleeding or a hereditary or acquired coagulation or platelet disorder), hepatic, immunological, renal, respiratory, genitourinary, or major neurological (including stroke, intercranial hemorrhage, and chronic seizures) abnormalities or diseases
* History of cancer (malignancy)

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-12-08 (Actual); Primary Completion 2026-04-12 (Estimated); Study Completion 2026-04-24 (Estimated)

PRIMARY OUTCOMES:
Area Under the Concentration-Time Curve from Time 0 to Infinity (AUC0-Inf) of Nemtabrutinib | Up to approximately 4 weeks
  Blood samples will be collected to determine the AUC0-inf of nemtabrutinib.
Maximum Plasma Concentration (Cmax) of Nemtabrutinib | Up to approximately 4 weeks
  Blood samples will be collected to determine the Cmax of nemtabrutinib.
Area Under the Concentration-Time Curve from Time 0 to Last (AUC0-Last) of Nemtabrutinib | Up to approximately 4 weeks
  Blood samples will be collected to determine the AUC0-last of nemtabrutinib.
Time to Maximum Plasma Concentration (Tmax) of Nemtabrutinib | Up to approximately 4 weeks
  Blood samples will be collected to determine the Tmax of nemtabrutinib.
Apparent Terminal Half-life (t1/2) of Nemtabrutinib | Up to approximately 4 weeks
  Blood samples will be collected to determine the t1/2 of nemtabrutinib.
Apparent Clearance (CL/F) of Nemtabrutinib | Up to approximately 4 weeks
  Blood samples will be collected to determine the CL/F of nemtabrutinib.
Volume of Distribution During Terminal Phase (Vz/F) of Nemtabrutinib | Up to approximately 4 weeks
  Blood samples will be collected to determine the Vz/F of nemtabrutinib.

SECONDARY OUTCOMES:
Number of Participants Who Experience an Adverse Event (AE) | Up to approximately 5 weeks
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. The number of participants who experience an AE will be reported.
Number of Participants Who Discontinue Study Treatment Due to an AE | Up to approximately 3 weeks
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. The number of participants who discontinue study treatment due to an AE will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (1):
- Fortea CRU Madison ( Site 0001), Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com/